CLINICAL TRIAL: NCT04279951
Title: Alpha and Omega of Lifestyle Therapy - Resistance Training and Ingestion of n-3 Polyunsaturated Fatty Acids to Improve Health and Muscle Functions in Individuals With Obesity and Healthy Controls
Brief Title: Alpha and Omega of Lifestyle Therapy
Acronym: Alpha&Omega
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Trainome 2019#015
Record Dates: First submitted 2020-01-19; First posted 2020-02-21 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Obesity
Keywords: Resistance exercise; Omega 3
MeSH Terms: conditions — Obesity | interventions — Resistance Training; Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Omega 3 (Experimental): Intake of 1 gram omega-3 (capsules) per day for 20 weeks
  + high-load and low-load resistance exercise two times per week for 10 weeks, preceded by 3 weeks of familiarization to training (high-load training)
  Interventions: Other: Resistance exercise; Dietary Supplement: Omega-3
- Placebo (Placebo Comparator): Intake of 1 gram sunflower oleic oil (capsules) per day for 20 weeks
  + high-load and low-load resistance exercise two times per week for 10 weeks, preceded by 3 weeks of familiarization to training (high-load training)
  Interventions: Other: Resistance exercise; Dietary Supplement: Placebo
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Resistance exercise — High-load and low-load resistance exercise two times per week for 10 weeks, preceded by 3 weeks of familiarization to training (high-load training)
  Arms: Omega 3; Placebo
Dietary Supplement: Omega-3 — 1 gram of omega-3 per day for 20 weeks
  Other Names: N-3 PUFA
  Arms: Omega 3
Dietary Supplement: Placebo — 1 gram of sunflower oleic oil per day for 20 weeks
  Arms: Placebo

SUMMARY:
The study aims to investigate the effects of double-blinded, randomized placebo-controlled n3-fatty acid supplementation (1000 mg day-1) and 13 weeks of resistance training on muscle function/biology and systemic health in individuals with obesity (BMI>30) and lean individuals (BMI<30)

DETAILED DESCRIPTION:
Lifestyle therapy is important for treating lifestyle-related morbidities such as obesity. Such therapy often includes exercise and nutrition, and leads to improved health, functionality and quality of life. Unfortunately, obesity leads to adverse changes in the physiological milieu, including inflammation and altered nutritional status such as reduced omega-3:omega-6 ratios. Indeed, inadequate omega 3 levels are common even among lean individuals. This may negatively affect the outcome of lifestyle therapy with exercise, particularly those involving resistance training, contributing to the large heterogeneity seen in training responses. In accordance with this, many individuals (including both lean and obese subjects) fail to improve muscle biology/functions and health, including failure to increase muscle mass and strength, failure to improve glucose handling and inflammatory status. This makes general lifestyle therapy recommendations ineffective. Here, we investigate effects of double-blinded, randomized placebo-controlled n3-fatty acid supplementation (1000 mg day-1) and 13 weeks of low- and high-load resistance training on muscle growth/function/biology and health in individuals with obesity (BMI>30, n=60) and lean controls (BMI<30, n=60). Each participant will perform two different training protocols, one on each leg. The supplement period will commence 7 weeks prior to the onset of the strength training intervention to ensure adequate omega-3 biology at the onset of training. Analyses include assessment of the separate and combined effects of n3-supplementation and obesity on training responses to resistance training, measured as muscle mass, muscle strength/functionality, muscle biological traits, and systemic health variables such as hormone/inflammation/glucose biology, adipose tissue biology/mass, gut microbiome and health-related quality of life. The project will provide important insight into the feasibility of resistance training and n-3 fatty acid supplementation for treating individuals with obesity, paving the way for personalized lifestyle therapy.

The study has two defined main outcome measures, targeting the combined effects of omega-3 and strength training on i) muscle thickness of the thigh (measured using ultrasound; this main outcome measure targets the effects of the intervention on muscle growth), and ii) glucose tolerance (measured using an oral glucose test; this main outcome measure targets the effects of the intervention on improvements in health).

In our analytical approach, we will use a mixed model-approach to assess the main effects of the intervention, mainly defined as changes from before to after the resistance training intervention. Importantly, for health variables such as glucose tolerance, analyses will be performed by accounting for individual variation at baseline, as any beneficial effect can be expected to be higher/present only in individuals with a pathological/diseased starting point. Notably, for many variables, we will collect data from two additional time points (pre-supplementation and after two weeks of familiarization to training). These data will provide insight into additional perspectives, such as the effects of omega-3 intake-only on glucose tolerance, which will bring additional depth to our conclusions (these analyses are not necessarily specified in the Outcome Measures section). For other data, such as primary cultivation of skeletal muscle and muscle mitochondrial respiration, data will only be collected from a randomized subset of participants. For analyses of the effects of the intervention on obesity-related pathophysiologies and health-related quality of life, data from a group of non-intervention individuals will act as reference values (data sampled alongside the intervention). Finally, we will use regression analyses to explain individual differences in training responses, with particular emphasis on muscle hypertrophy/glucose tolerance and their mechanistic origin of nature.

2021/08: The number of anticipated participants was increased from 120 to 150 due to circumstances relating to the SARS-CoV-2 pandemic

ELIGIBILITY:
Inclusion Criteria:

* Untrained (less than 2 sessions of resistance exercise per month and less than 3 hours of endurance exercise per week)

Exclusion Criteria:

* Unstable cardiovascular disease
* Injuries affecting the ability to perform heavy resistance exercise
* Mental illness
* Allergy to local anesthesia
* Smoking
* Use of medicine or drugs containing steroids the last two months prior to inclusion

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Muscle thickness, ultrasound | Changes from before to after the resistance training intervention (week 8 to 20)
  Muscle thickness of vastus lateralis and vastus intermedius measured using ultrasound
Glucose tolerance | Changes from before to after the resistance training intervention (week 8 to 20)
  Glucose tolerance measured using an oral glucose tolerance test

SECONDARY OUTCOMES:
Lean body mass | Changes from before to after the resistance training intervention (week 8 to 20)
  Lean body mass measured using whole-body DXA scan
Fat mass | Changes from before to after the resistance training intervention (week 8 to 20)
  Fat mass measured using whole-body DXA scan
Visceral fat mass | Changes from before to after the resistance training intervention (week 8 to 20)
  Visceral fat mass measured using whole-body DXA scan
Muscle mass, MRI | Changes from before to after the resistance training intervention (week 8 to 20)
  Thigh muscle cross sectional area/volume measured using magnetic resonance imaging (MRI)
Muscle mass, immunohistochemistry | Changes from before to after the resistance training intervention (week 8 to 20)
  Fibre type-specific muscle-fibre cross-sectional area measured using immunohistochemistry
Muscle mass, combined measure | Changes from before to after the resistance training intervention (week 8 to 20)
  Muscle mass of the legs measured as the weighted average of data from ultrasound, MRI, immunohistochemistry and DXA measurements
Muscle fibre type composition | Changes from before to after the resistance training intervention (week 8 to 20)
  Muscle fibre type composition measured using immunohistochemistry
Myonuclear number | Changes from before to after the resistance training intervention (week 8 to 20)
  Fiber type-specific myonuclear number measured using immunohistochemistry
Muscle satellite cell number | Changes throughout the course of the resistance training intervention (weeks 8, 10 and 20)
  Fiber type-specific muscle satellite cell number measured using immunohistochemistry
Muscle capillarization | Changes from before to after the resistance training intervention (week 8 to 20)
  Fiber type-specific muscle capillarization measured using immunohistochemistry
Fat infiltration (muscle) | Changes from before to after the resistance training intervention (week 8 to 20)
  Fat infiltration in thigh muscle measured using magnetic resonance imaging (MRI)
Muscle quality | Changes from before to after the resistance training intervention (week 8 to 20)
  Muscle strength measured per muscle mass of the legs
Unilateral lower body maximal strength | Changes throughout the course of the resistance training intervention (weeks 8, 10 and 20)
  The ability of muscles of the lower body to exert maximal force during dynamic movements
Unilateral lower body isokinetic muscle strength | Changes throughout the course of the resistance training intervention (weeks 8, 10 and 20)
  The ability of the knee extensors to exert maximal force during isokinetic movements
Unilateral lower body isometric muscle strength | Changes throughout the course of the resistance training intervention (weeks 8, 10 and 20)
  The ability of the knee extensors to exert maximal force during isometric actions
Peak power output during one-legged cycling | Changes from before to after the resistance training intervention (week 8 to 20)
  Maximal cycling performance measured as peak power output (Watt) during an incremental one-legged cycling test
Oxygen consumption during one-legged cycling | Changes from before to after the resistance training intervention (week 8 to 20)
  The ability to consume oxygen during an incremental one-legged cycling test
Unilateral lower body muscle endurance | Changes throughout the course of the resistance training intervention (weeks 8, 10 and 20)
  The ability of muscles of the lower body to perform repeated dynamic contractions at a specified submaximal load (70% of 1RM) to exhaustion
Waist circumference | Changes from before to after the resistance training intervention (week 8 to 20)
  Circumference of the waist measured using measuring tape
Blood pressure at rest | Changes from before to after the resistance training intervention (week 8 to 20)
  Blood pressure at rest measured using an automated upper-arm blood pressure cuff
Hemoglobin glycosylation (HbA1c) | Changes throughout the course of the intervention (weeks 0, 8 and 20)
  Long-term glucose levels measured as hemoglobin glycosylation of the metabolic syndrome such as waist circumference, blood pressure at rest, lipid profile ( hemoglobin glycosylation (HbA1c) and fasting blood glucose
Fasting blood glucose | Changes throughout the course of the intervention (weeks 0, 8 and 20)
  Fasting blood glucose measured in serum
N-3 PUFA (blood) | Changes throughout the course of the intervention (weeks 0, 8 and 20)
  Omega-3 (DHA/EPA) levels in blood
Inflammatory characteristics of peripheral blood mononuclear cell (PBMC) | Throughout the course of the intervention (weeks 0, 8 and 20)
  Expression of genes associated with inflammation and lipid metabolism in peripheral blood mononuclear cell measured using quantitative PCR
Lipid concentrations in blood | Changes throughout the course of the intervention (weeks 0, 8 and 20)
  Concentrations of various lipids and lipid metabolites such as triglycerides, LDL, HDL, ceramides, dihydroceramides, glucosylceramides, and lactosylceramides measured in serum using tageted metabolomics
Nutritent concentrations in blood | Changes throughout the course of the intervention (weeks 0, 8 and 20)
  Concentrations of nutrients (such as amino acids) and ions (such as iron and calcium) measured in serum
Hormone concentrations in blood | Changes throughout the course of the intervention (weeks 0, 8 and 20)
  Concentrations of hormones such as testosterone, growth hormone, thyroid hormones, cortisol and insulin (as well as c-peptide) measured in serum
Concentrations of inflammatory factors in blood | Changes throughout the course of the intervention (weeks 0, 8 and 20)
  Levels of inflammatory factors such as IL6, CRP and NFkB in serum
Muscle fractional synthesis rate | Week 18 to 20
  Protein/RNA synthesis rate measured using heavy water (deuterium) and chromatography/spectrometry
Gene expression in skeletal muscle (intervention) | Changes from before to after the resistance training intervention (week 8 to 20)
  RNA (e.g. messenger RNA, ribosomal RNA, microRNA, long non-coding RNA) abundances in m. vastus lateralis, measured both as targeted genes and at the level of the transcriptome
Gene expression in skeletal muscle (familiarization) | Changes from before to after familiarization to resistance exercise (week 8 to 10)
  RNA (e.g. messenger RNA, ribosomal RNA, microRNA, long non-coding RNA) abundances in m. vastus lateralis, measured both as single genes and at the level of the transcriptome
Protein abundance in skeletal muscle (intervention) | Changes from before to after the resistance training intervention (week 8 to 20)
  Levels of proteins and their modification status (e.g. phosphorylation) in m. vastus lateralis, measured at the level of single proteins and at the level of the proteome
Protein abundance in skeletal muscle (familiarization) | Changes from before to after the resistance training intervention (week 8 to 10)
  Levels of proteins and their modification status (e.g. phosphorylation) in m. vastus lateralis, measured at the level of single proteins and at the level of the proteome
Mitochondrial functions in muscle | Changes from before to after the resistance training intervention (week 8 to 20)
  The ability of muscle mitochondria (extracted from muscle homogenate) to synthesize ATP in vitro
Gene expression in subcutaneous fat | Changes from before to after the resistance training intervention (week 8 to 20)
  RNA (e.g. messenger RNA, ribosomal RNA, microRNA, long non-coding RNA) abundances in subcutaneous fat, measured as targeted genes
Satellite cell proliferation and myotube growth (in vitro) | Changes from before to after N3-supplementation-only (week 0 to 8)
  The ability of muscle satellite cells (extracted from muscle homogenate) to proliferate (rates of cell division), differentiate into myotubes and subsequently grow (rates of change in myotube size) in primary cultures
Musculoskeletal pain (Nordic Pain Questionnaire) | Changes throughout the course of the training intervention (weeks 0, 8 and 20)
  Musculoskeletal pain measured using The standardized Nordic Pain Questionnaire
Musculoskeletal pain (VAS) | Changes throughout the course of the training intervention (weeks 0, 8 and 20)
  Musculoskeletal pain measured using VAS-scale (1-10)
Gastrointestinal symptoms | Changes throughout the course of the training intervention (weeks 0, 8 and 20)
  Gastrointestinal symptoms such as abdominal discomfort and pain, measured using Rome IV criteria
Gut microbiome (feces, N3-supplementation-only) | Changes from before to after N3-supplementation-only (week 0 to 8)
  Relative composition of the gut microbiome measured using quantitative polymerase chain reaction
Gut microbiome (feces, training intervention) | Changes from before to after the resistance training intervention (week 8 to 20)
  Relative composition of the gut microbiome measured using quantitative polymerase chain reaction
Fecal short-chained fatty acids (N3-supplementation-only) | Changes from before to after N3-supplementation-only (week 0 to 8)
  Short chained fatty acids measured in feces
Fecal short-chained fatty acids (training intervention) | Changes from before to after the resistance training intervention (week 8 to 20)
  Short chained fatty acids measured in feces
Arterial stiffness | Throughout the course of the intervention (week 0, 8 and 20)
  Arterial stiffness measured using pulse-wave velocity
Health-related quality of life (SF-36) | Changes throughout the course of the intervention (week 0, 8 and 20)
  Health-related quality of life measured using the SF-36 questionnaire
Health-related quality of life in overweight/obesity | Changes throughout the course of the intervention (week 0, 8 and 20)
  Health-related quality of life in overweight/obesity individuals measured using The impact of weight on quality of life (IWQOL) questionnaire
Health-related quality of life (PANAS) | Changes throughout the course of the intervention (week 0, 8 and 20)
  Health-related quality of life measured using the Positive and Negative Affect Schedule (PANAS) questionnaire
Activities of daily living | Changes throughout the course of the intervention (week 0, 8 and 20)
  Activities of daily living (e.g. time spent in physical activity, intensities of activities) measured using questionnaire

OTHER OUTCOMES:
Training diary relating to the intervention protocol | Weeks 8 to 20
  Information about intervention-specific training, including training frequency, volume and load
Dietary registration | Week 0, 8 and 20
  Dietary registration measured using a food frequency questionnaire, assessing nutritional composition, energy intake and habitual patterns of dietary intake

CONTACTS AND LOCATIONS:
Overall Officials: Stian Ellefsen, PhD, Principal Investigator — Inland Norway University of Applied Sciences
Locations (1):
- Inland Norway University of Applied Sciences, Lillehammer, Norway